CLINICAL TRIAL: NCT02264353
Title: The Impact of Arousal Threshold in Obstructive Sleep Apnea: Donepezil's Effects on the Arousal Threshold and on the Apnea Hypopnea Index
Brief Title: The Impact of Arousal Threshold in Obstructive Sleep Apnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSD141272
Record Dates: First submitted 2014-09-17; First posted 2014-10-15 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive; Sleep Apnea; Arousal threshold; Donepezil
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Donepezil (Experimental): Sleep data with Donepezil given
  Interventions: Drug: Donepezil
- Placebo (Placebo Comparator): Sleep data with Placebo given
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Donepezil — Donepezil 10mg before sleep
  Arms: Donepezil
Drug: placebo — One piece of placebo before sleep
  Arms: Placebo

SUMMARY:
The investigators hypothesis is that obstructive sleep apnea (OSA) patients with a low arousal threshold may wake up too early during a respiratory event, before upper airway muscles can be activated to achieve stable ventilation. Thus, strategies to manipulate the respiratory arousal threshold could potentially improve the quality of sleep and sleep disordered breathing. Agents that raise arousal threshold are therefore likely to benefit some patients with OSA. The overall goal of this project is to determine the importance of the arousal threshold in OSA, determine which patients might benefit from a raised arousal threshold, and test this hypothesis by using pharmacological manipulation of the arousal threshold to achieve this goal.

DETAILED DESCRIPTION:
This study is a pilot study. The investigators will test whether donepezil has important effects on the arousal threshold and on the apnea hypopnea index.

Donepezil is a cholinesterase inhibitor approved by the U.S. Food and Drug Administration (FDA) for the treatment of symptoms of Alzheimer's disease.

Eligible participants will undergo overnight polysomonography as described below and will receive either donepezil (10 mg immediately prior to sleep) or placebo (in random order) followed roughly 14 days later with placebo or donepezil. This aim will allow us to test the impact of donepezil on the apnea hypopnea index. The study plans to enroll approximately 30 subjects.

The change in apnea hypopnea index as well as arousal thresholds/upper airway mechanics will be compared in the donepezil groups with the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 years
* sleep study (with apnea hypopnea index>5)
* Diagnosis of obstructive sleep apnea

Exclusion Criteria:

* Any known unstable cardiac (apart from treated hypertension), pulmonary (including asthma), renal, neurologic (including epilepsy), neuromuscular, or hepatic disease.
* Susceptible to stomach ulcers.
* Pregnant women or Nursing mothers
* Using positive airway pressure (PAP) therapy over one week or longer
* Body weight <55kg
* History of hypersensitivity to Afrin, Lidocaine and/or Donepezil
* History of bleeding diathesis and/or gastrointestinal bleeding.
* Use of any medications that may affect sleep or breathing.
* A psychiatric disorder, other than mild depression; e.g. schizophrenia, bipolar disorder, major depression, panic or anxiety disorders.
* Substantial cigarette (>5/day), alcohol (>3oz/day) or use of illicit drugs.
* More than 10 cups of beverages with caffeine (coffee, tea, soda/pop) per day.
* Deprived from sleep in the recent one week
* Desaturations to below 70% lasting greater than 10 seconds in duration per event in the sleep study (without Oxygen).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Owens, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Li Y, Orr J, Jen R, Sands SA, DeYoung P, Smales E, Edwards B, Owens RL, Malhotra A. Is there a threshold that triggers cortical arousals in obstructive sleep apnea. Sleep. 2019 Jun 11;42(6):zsz047. doi: 10.1093/sleep/zsz047. PMID 30794310
- [Derived] Li Y, Owens RL, Sands S, Orr J, Moraes W, DeYoung P, Smales E, Jen R, Malhotra A. The Effect of Donepezil on Arousal Threshold and Apnea-Hypopnea Index. A Randomized, Double-Blind, Cross-Over Study. Ann Am Thorac Soc. 2016 Nov;13(11):2012-2018. doi: 10.1513/AnnalsATS.201605-384OC. PMID 27442715

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil Then Placebo: Sleep data with Donepezil given during Visit 1 followed by a 14 day washout period followed by Sleep data with Placebo given during Visit 2
  Donepezil: Donepezil 10mg before sleep
- Placebo Then Donepezil: Sleep data with Placebo given during Visit 1 followed by a 14 day washout period followed by Sleep data with Donepezil given during Visit 2
  placebo: One piece of placebo before sleep
Period: Overall Study
Arm/Group | Donepezil Then Placebo | Placebo Then Donepezil
Started | 20 | 24
Completed | 17 | 24
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Donepezil 10mg tablet or Placebo tablet (matching Donepezil 10mg) before sleep
Arm/Group | All Study Participants
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 33
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41
Apnea Hypopnea Index (AHI)>5 events/hr; lowest Oxygen Saturation (SaO2)>70% [Count of Participants; unit: Participants] | 41

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI)
Description: The Apnea-Hypopnea Index or Apnoea-Hypopnoea Index (AHI) is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. The apneas (pauses in breathing) must last for at least 10 seconds and be associated with a decrease in blood oxygenation. A higher AHI value indicates more severe sleep apnea
Time Frame: 14 days (during overnight sleep study after donepezil or placebo is given)
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 41 | 41
events/hour | 50.0 (23.4) | 51.8 (27.4)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; Test type: Superiority; p = 0.576, t-test, 2 sided

2. Secondary Outcome: Respiratory Arousal Threshold
Description: Arousal Threshold was measured as the average nadir epiglottic airway pressure immediately before electroencephalogram (EEG) arousal. It was measured with an epiglottic pressure catheter. The epiglottic catheter/balloon is linked in a pressure catheter inserted through the de-congested, anesthetized nostril and the tip of the catheter located at hypopharyngeal area.
Time Frame: 14 days (during overnight sleep study after donepezil or placebo is given)
Measure: Mean (Full Range); unit: cm H20
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 21 | 21
cm H20 | -18.0 [-27.0 to -11.8] | -18.9 [-27.5 to -12.3]
Statistical Analysis 1: Comparison: Donepezil vs Placebo; Test type: Other; p = 0.394, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: Loop Gain
Description: The sensitivity of the ventilatory control system (loop gain) was quantified by fitting a simplified mathematical model to the spontaneous ventilatory pattern of obstructive sleep apnea (OSA). The sensitivity of the ventilatory control system (loop gain) was quantified by fitting a simplified mathematical model to the spontaneous ventilatory pattern of OSA 21. Loop gain is reflected in the size of the ventilatory overshoot following a ventilatory perturbation (hypopnea/apnea), where loop gain = response/disturbance. Ventilatory fluctuations are estimated using the square-root transformed nasal pressure waveform. Loop gain was reported as the ventilatory response to a 1 cycle/min disturbance (LG1); a value of LGn>1 yields periodic central apnea. Calculations were performed using MATLAB
Time Frame: 14 days (during overnight sleep study after donepezil or placebo is given)
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 41 | 41
Unitless | 0.55 (0.15) | 0.58 (0.16)
Statistical Analysis 1: Comparison: Donepezil vs Placebo; Test type: Superiority; p = 0.089, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Donepezil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 2/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=41) | Placebo (N=41)
Heart Burn (Investigations) | 0 (0) | 1 (1) — Subject reported "heart burn" and decided to quit after taking placebo.
Difficulty Falling Asleep (Investigations) | 0 (0) | 1 (1) — Subject reported difficulty falling asleep in laboratory after taking placebo.

LIMITATIONS AND CAVEATS:
Underlying mechanism(s) of sleep apnea is likely to vary across individuals such that one might predict that an intervention may only be effective in a subset of OSA patients. We did not measure upper airway gain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No